CLINICAL TRIAL: NCT02979301
Title: Low-Dose Tamoxifen to Reduce High Background Parenchymal Uptake on Molecular Breast Imaging
Brief Title: Impact of Low-dose Tamoxifen on BPU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carrie Hruska, Associate Professor, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB 16-008736
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-04

CONDITIONS: High Background Uptake on MBI
MeSH Terms: interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamoxifen 5 mg/day (Experimental): Women with high background uptake on MBI take 5 mg tam per day for 30 days.
  Interventions: Drug: Tamoxifen
- Tamoxifen 10 mg/day (Experimental): Women with high background uptake on MBI take 10 mg tam per day for 30 days.
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — 5 mg or 10 mg tamoxifen per day for 30 days.

SUMMARY:
The study will examine whether changes in background parenchymal uptake (BPU) on molecular breast imaging (MBI) can be induced by short-term use of low-dose tamoxifen. Women who have previously had high BPU on MBI will be recruited. Participants will take low-dose tamoxifen for a 30-day period, with post-tamoxifen MBI in order to investigate the impact of tamoxifen on BPU.

ELIGIBILITY:
Inclusion Criteria:The following are requirements for entry into the study:

1. Female, age 40 or older at the time of enrollment
2. Most recent MBI examination, performed within 3 years of enrollment, showed moderate or marked background parenchymal uptake
3. Mammogram performed within 12 months prior to enrollment that is available for comparison
4. Willing and able to return for MBI following 30 days of low-dose tamoxifen
5. If able to become pregnant

   1. Negative pregnancy test within 48 hours prior to study MBI exam(s)
   2. Agrees to avoid pregnancy during the study and for at least 2 months after study participation ends, by abstinence, barrier method, or nonhormonal contraception.
6. Understands and signs the consent form

   -

Exclusion Criteria:Subjects will be excluded if any of the following characteristics are present:

1) Evidence of suspected breast disease as defined by positive findings or recommendation for short-interval follow-up on most recent breast imaging (including mammography, MBI, MRI, ultrasound, etc.) not yet resolved prior to enrollment 2) Breast biopsy or breast surgery performed 6 months prior to enrollment 3) Bilateral breast implants or status post-bilateral prophylactic mastectomy 4) Pregnant or lactating 5) Current or recent use (within 6 months prior to enrollment) of any of the following drugs:

1. Systemic hormonal therapy (oral or transdermal patch formulations)
2. Hormonal contraception (oral, transdermal, implanted, or injected formulations)
3. Selective estrogen receptor modulators (tamoxifen, raloxifene, or toremifene)
4. Aromatase inhibitors (anastrazole, letrozole, or exemestane)
5. GnRH analogs
6. Prolactin inhibitors
7. Androgens or antiandrogens
8. Anticoagulants or "blood thinners" (warfarin, heparin, rivaroxaban and other novel anticoagulants)
9. Drugs known to be strong inhibitors of CYP2D6, the major P450 enzyme that metabolizes tamoxifen, including:

   * bupropion (Wellbutrin)
   * fluoxetine (Prozac)
   * paroxetine (Paxil)
   * quinidine (Quinidex) 6) Personal history of any type of malignancy, with the exclusion of non-melanoma skin cancer, diagnosed prior to enrollment 7) Personal history or strong family history of blood clots in legs or lungs (also known as deep vein thrombosis or pulmonary embolism) 8) Personal history of transient ischemic attack (TIA) or cerebrovascular accident (CVA) 9) Active proliferative disorders of the endometrium such as atypical hyperplasia, history of active endometriosis, unresected polyps 10) Any type of retinal disorders or severe cataract 11) Current or former smoker 12) Known carrier of BRCA1 or BRCA2 genetic mutation or known DNA repair defect.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Hruska, PhD R-D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Hruska CB, Hunt KN, Conners AL, Geske JR, Brandt KR, Degnim AC, Vachon CM, O'Connor MK, Rhodes DJ. Impact of short-term low-dose tamoxifen on molecular breast imaging background parenchymal uptake: a pilot study. Breast Cancer Res. 2019 Mar 8;21(1):38. doi: 10.1186/s13058-019-1120-5. PMID 30850011
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Tamoxifen 5 mg/Day: Women with a history of high background uptake on MBI were enrolled.
  A baseline MBI was performed at Day 0. Women then took 5 mg tamoxifen per day for 30 days, followed by a post-tamoxifen MBI exam.
- Tamoxifen 10 mg/Day: Women with a history of high background uptake on MBI were enrolled.
  A baseline MBI was performed at Day 0. Women then took 10 mg tamoxifen per day for 30 days, followed by a post-tamoxifen MBI exam.
Period: Overall Study
Arm/Group | Tamoxifen 5 mg/Day | Tamoxifen 10 mg/Day
Started | 11 | 11
Completed | 10 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamoxifen 5 mg/Day | Tamoxifen 10 mg/Day | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (4.4) | 48.1 (4.0) | 47.7 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Background Parenchymal Uptake (BPU) on Molecular Breast Imaging (MBI)
Description: An image analysis tool to obtain a quantitative measure of background parenchymal uptake (BPU) was applied to pre-tamoxifen and post-tamoxifen MBI exams. The percent change in BPU from pre-tamoxifen to post-tamoxifen MBI was determined.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: percent change in BPU
Arm/Group | Tamoxifen 5 mg/Day | Tamoxifen 10 mg/Day
Number analyzed (Participants) | 10 | 11
percent change in BPU | 0.0 (21) | -12 (11)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until the last study visit for each study subject, approximately 30 days
Arm/Group | Tamoxifen 5 mg/Day | Tamoxifen 10 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT02979301/Prot_SAP_000.pdf